CLINICAL TRIAL: NCT04042961
Title: Effect of Reactive Balance Training on Physical Fitness Post-stroke
Brief Title: Reactive Balance Training and Fitness
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: University of Toronto (Other); Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Avril Mansfield, Principal Investigator, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-5784
Record Dates: First submitted 2019-07-29; First posted 2019-08-02 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: CVA (Cerebrovascular Accident)
MeSH Terms: conditions — Stroke | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reactive balance training (Experimental)
  Interventions: Other: Reactive balance training
- Aerobic and strength training (Active Comparator)
  Interventions: Other: Aerobic and strength training (AST)

INTERVENTIONS:
Other: Reactive balance training — A variety of tasks will be included to induce external or internal perturbations. External perturbations will be caused by forces outside participants' control (e.g. a push or pull from the physiotherapist). Internal perturbations are when the participant fails to control the centre of mass-base of support relationship during voluntary movement; e.g., 'agility' tasks such as kicking a soccer ball. Each session will include a five-minute warm-up, at least 60 perturbations, and a five-minute cool-down. The difficulty of the task will be set such that participants will 'fail' to recover balance ~50% of the time; 'failure' is defined as use of an upper extremity response, use of external assistance (i.e. from the overhead harness or physiotherapist), or taking more than 2 steps to regain stability. Training tasks will progressed by increasing the perturbation magnitude, including cognitive or movement tasks, or imposing sensory or environmental challenges (e.g. eyes closed, obstacles).
  Arms: Reactive balance training
Other: Aerobic and strength training (AST) — AST sessions will consist of 30 minutes of aerobic and 30 minutes of strength training.
  Aerobic training: Aerobic training will be done using treadmill walking or combination of modalities (e.g. cycling or recumbent stepping) for those unable to maintain the target heart rate with walking. The heart rate that occurred at the ventilatory threshold (V̇O2VT) during the cardiopulmonary exercise test will be used to prescribe intensity. In the absence of a discernible V̇O2VT a combination of the following will be used: 60-80% of heart rate reserve, peak oxygen uptake, and rating of perceived exertion of 11-16 (Borg 6-20 scale). Prescriptions will be initially progressed by increasing duration to ≥20 minutes and then increasing intensity to target heart rate.
  Resistance training: Participants will be prescribed 1-2 sets of 8 exercises per session (squat, heel raise, ankle dorsiflexion, knee extension and flexion, abdominal curl-up, wall push up, bicep curl), at 70% of 1 repetition maximum.
  Arms: Aerobic and strength training

SUMMARY:
People with stroke should exercise to maintain function and reduce the risk of another stroke. Different types of exercise target different components of fitness, such as aerobic, strength, and balance. Post-stroke exercise guidelines exist for each type of exercise separately (eg, brisk walking as aerobic exercise, resistance training for strength, and Tai Chi for balance). Meeting these recommendations means spending a lot of time exercising, and people with stroke say that lack of time and fatigue are barriers to exercise. It is possible to target several components of fitness with one type of exercise.

'Reactive balance training' (RBT) is a type of exercise that improves control of reactions that are needed to prevent a fall after losing balance, and is the only type of exercise with potential to prevent falls in daily life post-stroke. Because RBT involves repeated whole-body movements it may have similar aerobic benefit as other exercises using whole-body movements (eg, brisk walking). Also, leg muscles need to generate a lot of force to make rapid steps in RBT; repeatedly generating this force may help to improve strength.

The purpose of this study is to determine if RBT improves two important components of fitness among people with chronic stroke: aerobic capacity and strength. The investigators expect that the improvements in aerobic capacity and strength after RBT will not be any worse than after an exercise program that specifically targets aerobic fitness and strength. A secondary purpose of this study is to determine the effects of RBT compared to aerobic and strength training on balance control and balance confidence. The investigators expect that RBT will lead to greater improvements in balance control and balance confidence than an aerobic and strength training program.

DETAILED DESCRIPTION:
This is an assessor-blind randomized non-inferiority trial with an internal pilot study. Research activities will take place at the Toronto Rehabilitation Institute and the University of Toronto. For the internal pilot study, we will initially recruit 20 participants with chronic stroke and randomly assign them to one of two groups: 1) RBT, or 2) AST. Cardiorespiratory fitness, lower-extremity strength, balance control, and balance confidence will be measured pre- and post-intervention. We will calculate the final target sample size using the variability observed in this internal pilot. Additionally, a Trial Steering Committee will determine the criteria for the progression from the internal pilot to the main study, and will decide on the continuation of the internal pilot with or without modifications based on those pre-defined criteria (e.g., criteria based on feasibility or preliminary evidence of effect of the interventions from examination of effect sizes).

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults with chronic stroke (>6 months post-stroke).
* Able to stand independently without upper-limb support for >30 seconds.
* Able to tolerate at least 10 postural perturbations while wearing a safety harness.

Exclusion Criteria:

* >2.1m tall and/or weighing >150kg (limits of the safety harness system).
* Other neurological condition that could affect balance control (e.g., Parkinson's disease).
* Lower extremity amputation.
* Cognitive, language or communication impairments affecting understanding instructions.
* Recent (last 6 months) significant illness, injury or surgery.
* Severe osteoporosis, defined by diagnosis of osteoporosis with fracture.
* Severe uncontrolled hypertension, or uncontrolled diabetes.
* Contraindications to exercise testing, such as symptomatic aortic stenosis, complex life-threatening arrhythmias, unstable angina, or orthostatic blood pressure decrease of >20 mmHg with symptoms.
* Acute or chronic illness or injury likely to be exacerbated by exercise (e.g., recent lower-extremity fracture).
* Currently attending in- or out-patient physiotherapy, in which they receive aerobic training, balance training or strength training for lower limb.
* Significant exercise participation: current physical activity levels that meet the recommended guidelines (at least 150 minutes of moderate-to-vigorous or at least 75 minutes of vigorous physical activity/week) as calculated using the moderate and vigorous components of the Leisure Time Exercise Questionnaire (LTEQ) in the month prior to starting the study.
* Received perturbation training at Toronto Rehab <1 year previously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Aerobic capacity | Data will be collected immediately pre- and post-intervention. We will analyse the change in the outcome from pre- to post-intervention.
  A symptom-limited cardiopulmonary exercise test (CPET) will be performed. The CPET will be medically supervised. It will be conducted on the same modality on subsequent assessments and at the same time of day as the supervised exercise classes to minimize effects of heart rate altering medication on exercise prescription. Resistance will be increased every minute until either the patient indicates that he/she would like to stop or abnormalities appear that necessitate discontinuing the test. Breath-by-breath gas samples will be collected via calibrated metabolic cart to determine V̇O2peak and V̇O2VT.
Lower extremity strength | Data will be collected immediately pre- and post-intervention. We will analyse the change in the outcome from pre- to post-intervention.
  Peak isokinetic torque will be measured using a isokinetic dynamometer. Participants will be seated in the chair (hips at approximately 90 degrees) with the axis of rotation of the dynamometer aligned to the femoral condyles. Shoulder straps will secure the torso and a thigh strap over the active leg will minimize compensatory movements during testing. The inactive leg will be positioned at 90 degrees knee flexion and held in place with a padded bar below the seat. Peak isokinetic muscle torque at a speed of 60 degrees/s will be assessed. Two to three warm-up contractions will be performed at ~50-75% of perceived maximum effort. This will be followed by 5 maximal efforts to obtain peak torque. A one-minute rest will be given between trials to minimize fatigue. The highest torque achieved among the three maximal trials will be used as the peak isokinetic torque. The task will be performed for both legs.

SECONDARY OUTCOMES:
Berg balance scale | Data will be collected immediately pre- and post-intervention. We will analyse the change in the outcome from pre- to post-intervention.
  Construct: Functional balance Scale range: 0-56 Higher values represent improved outcome
Mini-Balance Evaluation Systems Test | Data will be collected immediately pre- and post-intervention. We will analyse the change in the outcome from pre- to post-intervention.
  Construct: Anticipatory balance control, reactive balance control, gait, and sensory orientation in balance Scale range: 0-28 (total), 0-6 (anticipatory balance control), 0-6 (reactive balance control), 0-10 (gait), 0-6 (sensory orientation) Higher values represent improved outcome The total score is created by adding the sub-scale scores
Six-minute walk test | Data will be collected immediately pre- and post-intervention. We will analyse the change in the outcome from pre- to post-intervention.
Activities-specific Balance Confidence scale | Data will be collected immediately pre- and post-intervention. We will analyse the change in the outcome from pre- to post-intervention.
  Construct: balance confidence Scale range: 0-100 Higher values represent improved outcome
Falls in daily life | For 12 months post-intervention
  A fall is defined as "an event that results in a person coming to rest unintentionally on the ground or other lower level". Participants will complete a 12-month falls monitoring period after completing the initial training period. Participants will be provided stamped address postcards containing a calendar to record falls, which they will complete daily. Participants will return each postcard to the research team fortnightly. If a participant does not complete the event tracking within two weeks the research assistant will call them. In this telephone call, the research assistant will try to ascertain if the participant has experienced a fall in the previous two weeks. Participants who report a fall on the calendar will be contacted by the to complete a questionnaire asking about the circumstances of the fall.
Physical Activity Scale for Individuals with Physical Disabilities | 4 months, 8 months, and 12 months post-intervention
  Construct: physical activity in daily life Scale range: not applicable (the maximum score that is technically achievable would not be feasible) Higher scores represent improved outcome
Subjective Index of Physical and Social Outcome | 4 months, 8 months, and 12 months post-intervention
  Construct: participation Scale range: 0-40 (total); 0-20 (social sub-scale), 0-20 (physical sub-scale) Higher scores represent improved outcome The total score is the sum of the sub-scale scores

CONTACTS AND LOCATIONS:
Overall Officials: Avril Mansfield, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mansfield A, Aqui A, Danells CJ, Knorr S, Centen A, DePaul VG, Schinkel-Ivy A, Brooks D, Inness EL, Mochizuki G. Does perturbation-based balance training prevent falls among individuals with chronic stroke? A randomised controlled trial. BMJ Open. 2018 Aug 17;8(8):e021510. doi: 10.1136/bmjopen-2018-021510. PMID 30121600
- [Background] Marzolini S, Brooks D, Oh P, Jagroop D, MacIntosh BJ, Anderson ND, Alter D, Corbett D. Aerobic With Resistance Training or Aerobic Training Alone Poststroke: A Secondary Analysis From a Randomized Clinical Trial. Neurorehabil Neural Repair. 2018 Mar;32(3):209-222. doi: 10.1177/1545968318765692. Epub 2018 Mar 30. PMID 29600726
- [Background] Boyne P, Reisman D, Brian M, Barney B, Franke A, Carl D, Khoury J, Dunning K. Ventilatory threshold may be a more specific measure of aerobic capacity than peak oxygen consumption rate in persons with stroke. Top Stroke Rehabil. 2017 Mar;24(2):149-157. doi: 10.1080/10749357.2016.1209831. Epub 2016 Jul 25. PMID 27454553
- [Background] Flansbjer UB, Holmback AM, Downham D, Lexell J. What change in isokinetic knee muscle strength can be detected in men and women with hemiparesis after stroke? Clin Rehabil. 2005 Aug;19(5):514-22. doi: 10.1191/0269215505cr854oa. PMID 16119407
- [Derived] Barzideh A, Marzolini S, Danells C, Jagroop D, Huntley AH, Inness EL, Mathur S, Mochizuki G, Oh P, Mansfield A. Effect of reactive balance training on physical fitness poststroke: study protocol for a randomised non-inferiority trial. BMJ Open. 2020 Jun 30;10(6):e035740. doi: 10.1136/bmjopen-2019-035740. PMID 32606059